CLINICAL TRIAL: NCT00861861
Title: Comparison of Pitavastatin With Atorvastatin in Increasing HDL-C and Adiponectin in Patients With Dyslipidemia and Coronary Artery Disease.
Brief Title: Comparison of Pitavastatin With Atorvastatin in Increasing High Density Lipoprotein - Cholesterol (HDL-C) and Adiponectin in Patients With Dyslipidemia and Coronary Artery Disease (CAD)
Acronym: COMPACT-CAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kumamoto University (Other)
Responsible Party: Principal Investigator, Hisao Ogawa, Kumamoto University, Kumamoto University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kumamoto-746
Record Dates: First submitted 2009-03-12; First posted 2009-03-16 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Hypercholesterolemia; Coronary Artery Disease
Keywords: Pitavastatin; Atorvastatin; CAD; HDL-C; Adiponectin
MeSH Terms: conditions — Hypercholesterolemia; Coronary Artery Disease | interventions — pitavastatin; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): pitavastatin group
  Interventions: Drug: Pitavastatin
- 2 (Active Comparator): atorvastatin group
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Pitavastatin — comparison of two drugs in increasing HDL-C and adiponectin
  Arms: 1
Drug: Atorvastatin — comparison of two drugs in increasing HDL-C and adiponectin
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effects of pitavastatin and atorvastatin on adiponectin percentage change in patients with hypercholesteremia comorbid stable CAD.

DETAILED DESCRIPTION:
The efficiency of lipid lowering therapy was already proven by the clinical trials of statins. According to these results, the target value of LDL-C is recommended under 100mg/dL in the Japan Atherosclerosis Society Guidelines. However, the efficiency of intensive therapy to lower LDL-C more than 100mg/dL has not been proven yet.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dyslipidemia as defined by any of the parameters:

  * HDL-C < 50 mg/dL
  * LDL-C ≥ 140 mg/dL
  * LDL-C ≥ 100 mg/dL and cholesterol-lowering treatment is necessary in accordance with the investigator's judgement
* Patients who passed three months or more after acute myocardial infarction
* Patients who passed one month or more after unstable angina
* Patients who passed one month or more after PCI
* Patients with written consent by their own volition after being provided sufficient explanation for the participation into this clinical trial

Exclusion Criteria:

* Patients with any allergy to pitavastatin or atorvastatin
* Patients with familial hypercholesterolemia
* Patients receiving pitavastatin
* Patients with severe hypertension
* Patients with renal disorders or undergoing dialysis
* Patients with hepatobiliary disorders
* Patients with hepatobiliary disorders
* Patients with family history of hypothyroidism or muscular dystrophy
* Patients with history of drug-induced hepatic disorder
* Drug abuser or dipsomaniac
* Patients with cardiogenic shock.
* Patients who hopes for pregnancy during this study
* Contraindications, Relative Contraindications, Absolute Contraindications for Coadministration and Relative Contraindications for Coadministration for pitavastatin or atorvastatin
* Patients who are ineligible in the opinion of the investigator

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2008-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
HDL-cholesterol (HDL-C); Adiponectin; High-Molecular- Weight Adiponectin(HMW Adiponectin) | start, 6 months, 12 months, 30 months

SECONDARY OUTCOMES:
TC; LDL-C; HDL-C; HDL2-C; HDL3-C; TG; smalldenseLDL; MDA-LDL; FPG; HbA1c; Cr; RLP-C; apoA-I; apoB; apoC-Ⅱ; apoC-Ⅲ | start, 6 months, 12 months, 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Hisao Ogawa, MD,PhD, Principal Investigator — Kumamoto University Graduate School of Medical Sciences
Locations (1):
- Kumamoto University Graduate School of Medical Sciences Department of Cardiocascular Medicine, Kumamoto, Kumamoto, Japan